CLINICAL TRIAL: NCT04999293
Title: Antiplatelet Therapy in Elderly Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Ticagrelor in Elderly Patients Undergoing Percutaneous Coronary Intervention
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Meng Shaoke, M.D., The First Affiliated Hospital of Dalian Medical University
Other Study IDs: PJ-KS-KY-2021-146
Record Dates: First submitted 2021-08-05; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Platelet Aggregation Inhibitors; Dual Anti-Platelet Therapy; Aged; Percutaneous Coronary Intervention
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The Elderly Undergoing Percutaneous Coronary Intervention: Patients were survivors and treated with DAPT (aspirin [100 mg once daily], cilostazol, or indobufen)combined with a P2Y12 receptor antagonist [clopidogrel (75 mg once daily) or ticagrelor (90 mg twice daily)]) at the time of hospital discharge.All patients were followed for 1 year in the outpatient clinic after hospital discharge.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — Patients were survivors and treated with DAPT (aspirin [100 mg once daily], cilostazol, or indobufen)combined with a P2Y12 receptor antagonist [clopidogrel (75 mg once daily) or ticagrelor (90 mg twice daily)]) at the time of hospital discharge.All patients were followed for 1 year in the outpatient clinic after hospital discharge.
  Other Names: Clopidogrel

SUMMARY:
The study is an investigator-sponsored, retrospective cohort study designed to compare efficacy and safety of ticagrelor in elderly patients undergoing percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age≥75 years old;
* Treated with PCI (limited to stent implantation) ;
* Survivors and treated with DAPT (aspirin [100 mg once daily], cilostazol, or indobufen)combined with a P2Y12 receptor antagonist [clopidogrel (75 mg once daily) or ticagrelor (90 mg twice daily)]) at discharge;

Exclusion Criteria:

* Coronary artery bypass graft (CABG) or only drug conservative treatment during hospitalization;
* Concurrent use of oral anticoagulants;
* Inability to tolerate long-term antiplatelet therapy, such as active bleeding and a bleeding tendency;
* Acute infectious diseases;
* Cognitive impairment;
* Declined re-examination.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients ≥75 years of age who were treated with PCI (limited to stent implantation) at the First Affiliated Hospital of Dalian Medical University from January 1, 2015 to December 31, 2019 were screened for additional enrollment criteria.
Sampling Method: Probability Sample
Enrollment: 1505 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Types 2, 3, and 5 bleeding, as defined by the Bleeding Academic Research Consortium | 12 months
  The primary safety endpoint
Combined major adverse cardiovascular and cerebrovascular events (MACCEs), including all-cause mortality, myocardial infarction, ischemic stroke, and any revascularization. | 12 months
  The primary efficacy endpoint

SECONDARY OUTCOMES:
All-cause mortality | 12 months
Myocardial infarction | 12 months
Revascularization | 12 months
Ischemic stroke | 12 months
Incidence of BARC3 and 5 bleeding | 12 months
Incidence of major and minor bleeding defined by the PLATO study | 12 months
Incidence of major and minor bleeding defined by the TIMI study | 12 months
Occurrence of any bleeding | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shaoke Meng, MD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mehta SR, Yusuf S, Peters RJ, Bertrand ME, Lewis BS, Natarajan MK, Malmberg K, Rupprecht H, Zhao F, Chrolavicius S, Copland I, Fox KA; Clopidogrel in Unstable angina to prevent Recurrent Events trial (CURE) Investigators. Effects of pretreatment with clopidogrel and aspirin followed by long-term therapy in patients undergoing percutaneous coronary intervention: the PCI-CURE study. Lancet. 2001 Aug 18;358(9281):527-33. doi: 10.1016/s0140-6736(01)05701-4. PMID 11520521
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Husted S, James S, Becker RC, Horrow J, Katus H, Storey RF, Cannon CP, Heras M, Lopes RD, Morais J, Mahaffey KW, Bach RG, Wojdyla D, Wallentin L; PLATO study group. Ticagrelor versus clopidogrel in elderly patients with acute coronary syndromes: a substudy from the prospective randomized PLATelet inhibition and patient Outcomes (PLATO) trial. Circ Cardiovasc Qual Outcomes. 2012 Sep 1;5(5):680-8. doi: 10.1161/CIRCOUTCOMES.111.964395. PMID 22991347
- [Background] Gimbel M, Qaderdan K, Willemsen L, Hermanides R, Bergmeijer T, de Vrey E, Heestermans T, Tjon Joe Gin M, Waalewijn R, Hofma S, den Hartog F, Jukema W, von Birgelen C, Voskuil M, Kelder J, Deneer V, Ten Berg J. Clopidogrel versus ticagrelor or prasugrel in patients aged 70 years or older with non-ST-elevation acute coronary syndrome (POPular AGE): the randomised, open-label, non-inferiority trial. Lancet. 2020 Apr 25;395(10233):1374-1381. doi: 10.1016/S0140-6736(20)30325-1. PMID 32334703
- [Derived] Meng S, Guo L, Ye Z, Wang J, Ding H, Wu S, Huang R. Comparison of Clinical Outcomes Between Ticagrelor and Clopidogrel in Elderly Patients Undergoing Percutaneous Coronary Intervention: A Cohort Study. Clin Interv Aging. 2022 Apr 2;17:331-341. doi: 10.2147/CIA.S355210. eCollection 2022. PMID 35400997